CLINICAL TRIAL: NCT03381118
Title: A Randomized Study of Haploidentical Lymphocytes With Nivolumab and Intermediate Dose Cytarabine Versus Nivolumab and Intermediate Dose Cytarabine as Consolidation Treatment in Older Adults With Acute Myeloid Leukemia.
Brief Title: Haploidentical Lymphocytes With Nivolumab/Ara-C as Consolidation in Elderly AML Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unexpected toxicity
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 31/17-n
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ara-C+HaploLymphocyte+Nivo (Experimental): Patients treated with nivolumab, intermediate dose cytarabine and haploidentical lymphocyte infusion:
  [Cytarabine 500-1000 mg/m2 bid D-4, -3, -2 + G-CSF mobilized HLA-haploidentical donor peripheral blood stem cells infusion D0
  + Nivolumab 40 mg D+5] х 2-3 cycles
  Interventions: Drug: Cytarabine; Drug: Nivolumab; Biological: G-CSF mobilized HLA-haploidentical donor PBSC
- Ara-C+ Nivo (Experimental): Patients treated with nivolumab and intermediate dose cytarabine:
  [Cytarabine 500-1000 mg/m2 bid D+1, +2, +3 + Nivolumab 40 mg D+1] х 2-3 cycles
  Interventions: Drug: Cytarabine; Drug: Nivolumab

INTERVENTIONS:
Drug: Cytarabine — Cytarabine 500-1000 mg/m2 bid IV infusion on D-4, -3, -2
  Other Names: Ara-C
  Arms: Ara-C+HaploLymphocyte+Nivo
Drug: Nivolumab — Nivolumab 40 mg IV infusion on D+5
  Other Names: Opdivo
  Arms: Ara-C+HaploLymphocyte+Nivo
Drug: Cytarabine — Cytarabine 500-1000 mg/m2 bid IV infusion on D+1, +2, +3
  Other Names: Ara-C
  Arms: Ara-C+ Nivo
Drug: Nivolumab — Nivolumab 40 mg IV infusion on D+1
  Other Names: Opdivo
  Arms: Ara-C+ Nivo
Biological: G-CSF mobilized HLA-haploidentical donor PBSC — G-CSF mobilized HLA-haploidentical donor peripheral blood stem cells IV infusion on D0
  Arms: Ara-C+HaploLymphocyte+Nivo

SUMMARY:
A phase II trial to compare the efficacy and safety of nivolumab and intermediate dose cytarabine with or without haploidentical lymphocyte infusion. To identify the role of haploidentical lymphocytes in the treatment of acute myeloid leukemia in older adults. The patients will be stratified based on the remission number (first or second)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of acute myeloid leukemia with the confirmed first or second complete remission
* ≥ 55 years of age
* Not candidates for allogeneic stem cell transplantation as decided by the panel of hematologists at the transplant center
* Patients with a HLA-haploidentical donor who should be able to provide informed consent for peripheral blood apheresis
* No severe concurrent illness that limits life expectancy to less than 2 years

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Karnofsky index <70%
* Acute promyelocytic leukemia
* Other tumor requiring treatment at the time of enrollment
* Active or prior documented autoimmune disease requiring systemic treatment
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  DFS will be assessed with Kaplan-Meier method from the date of last remission before randomization until the date of relapse or the date of death

SECONDARY OUTCOMES:
Overall survival | 2 years
  OS will be assessed with Kaplan-Meier method from the date of last remission before randomization until the date of death from any cause
Incidence of graft-versus-host disease | up to 12 months
  Incidence of acute GVHD, grades I-IV
Treatment-related adverse events as assessed by CTCAE v4.03 | up to 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).

CONTACTS AND LOCATIONS:
Locations (1):
- Boris V Afanasyev, MD, Prof., Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided